CLINICAL TRIAL: NCT04880772
Title: A Single-centre Two-armed Randomised Controlled Trial Comparing Standard Care Alone Versus Exercise and Nutrition Prehabilitation in Elective Patients Undergoing Resectional HPB and Colorectal Cancer Surgery
Brief Title: Clinical Trial Comparing Standard Care Versus Prehabilitation in Patients Undergoing Cancer Surgery
Acronym: SPECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Lancashire Hospitals NHS Trust (Other)
Collaborators: Lancaster University (Other)
Responsible Party: Principal Investigator, Joel Lambert, Clinical Research Fellow, East Lancashire Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 290723
Record Dates: First submitted 2021-04-27; First posted 2021-05-11 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Cancer of Colon; Cancer of Rectum; Liver Metastases
Keywords: prehabilitation; surgery; cardiopulmonary exercise testing; cytokines
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation to standard care or prehabilitation
Who Masked: Outcomes Assessor
Masking Description: CPET clinician/physiologist will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Standard Care: Surgery school as per ELHT pre-operative guidelines (includes generic pre-operative information, advice and optimisation e.g correction of anaemia)
- Prehabilitation (Experimental): Surgery School plus Moderate intensity exercise & Forceval (multivitamin)
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — exercise & multivitamin (nutritional/dietary advice)
  Arms: Prehabilitation

SUMMARY:
To determine whether exercise and nutrition prehabilitation improves patient outcomes after cancer surgery

DETAILED DESCRIPTION:
Preliminary qualitative and quantitative studies suggest that there are benefits (reduced length of stay, improved cardiorespiratory function, reduced postoperative complications and improved quality of life) when prehabilitation is used with the context of cancer care. In 2017 Macmillian Cancer Support developed a strategic 'Evidence and Insight' review on prehabilitation. The outcome of this was to incorporate prehabilitation into routine cancer care and to develop principles and guidance for prehabilitation. This study aims to support this vision and answer some of the questions on the patients who are most likely to benefit from prehabilitation and to quantify some of these benefits by investigating the molecular processes that influence clinical changes

This study primarily seeks to assess the cardiovascular and biological impact of prehabilitation (exercise, nutrition) on patients undergoing hepatobiliary and colorectal cancer surgery. The investigators aim to assess whether there is an improvement in various cardiopulmonary exercise testing (CPET) variables such as maximum oxygen consumption and anaerobic threshold. The investigators also aim to study the inflammatory cytokines associated with cancer and how these markers respond to exercise. These inflammatory markers are thought to play a role in influencing some clinical outcomes such as wound infection and recovery.

The study will also assess secondary outcomes including hospital stay, post operative complications and quality of life. The investigators aim to better understand the biological relationship between anti-inflammatory cytokine levels and the previously mentioned outcomes by measuring and analysing these mediators and performing selected muscle biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85
* Sex: male/female
* Radiological/tissue cancer diagnosis
* Curative cancer of the colon, rectum, colorectal liver metastases (CRLM) of 2 or more segments
* elective surgery (planned a minimum of 3 weeks from the date of first clinic meeting)
* Access to digital technology(mobile phone, tablet or laptop, home computer) to participate in supervised home exercise

Exclusion Criteria:

Exclusion

* Palliative disease
* Haematological malignancy
* Pregnancy
* Emergency surgery
* Physically unable to undergo CPET
* Part of any other trial with similar interventions unless previously agreed on with all CIs
* synchronous disease (operation on HPB & colorectal cancers at the same operation)
* No access to digital technology(smart phone, tablet, laptop or home computer)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Anaerobic threshold (AT) measured in ml/kg/min and maximum oxygen consumption ( VO2 peak) measured in ml/kg/min | change in baseline AT & VO2 peak at 4 weeks
  Cardiopulmonary exercise Test (CPET) variables
Inflammatory cytokines | change in baseline cytokines at 4 weeks
  IL6 IL10 in muscle and blood measured in pg/ml

SECONDARY OUTCOMES:
Clavien-Dindo complication rates | Up to 30 days from the day of operation
  Grades I-IV
Length of hospital stay measured in days | 30 & 90-day mortality
  Defined as duration of stay from date of operation to discharge
Quality of life measures (Illness Perception Questionnaire) | baseline and within 24 weeks after surgery
  This questionnaire assesses perceptions on each of the five dimensions(Identity, Cause, Timeline, Consequences, Cure-Control) by asking patients for their own beliefs about their condition.
  High scores on the identity, consequences, timeline acute/ chronic and cyclical subscales represent strongly held beliefs about the number of symptoms attributed, the negative consequences, and the chronicity and cyclical nature of the illness.
  High scores on the identity and cure-control and coherence subscales represent positive beliefs about controllability and a personal understanding of the illness.
Hand Grip Strength measured in kg | baseline, immediately after the intervention, within 24 weeks after surgery
  Measured by digital dynamometer
Quality of life measure (Mental Adjustment to Cancer Scale) | baseline and within 24 weeks after surgery
  Assessment of participants mental adjustment to a cancer diagnosis. Designed to measure Fighting Spirit (FS), Anxious Preoccupation (AP), Helpless-hopelessness (HH) and Fatalism. This is a 40-item measure of specific psychological (Coping) responses that cancer patients may display in the process of adjusting to the diagnosis and treatment of their disease.
  A higher score represents higher endorsement of the adjustment response.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Lambert, Principal Investigator — Senior Clinical Research Fellow; Chris Gaffney, Study Director — Lancaster University
Locations (1):
- Royal Blackburn Hospital, Blackburn, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised CPET data to be shared with other researchers. Anonymised tissue and blood samples to be shared with other researchers for analysis
Supporting Information: Study Protocol, SAP
Time Frame: 18 months
Access Criteria: Full anonymisation

REFERENCES:
- [Background] Lambert JE, Hayes LD, Keegan TJ, Subar DA, Gaffney CJ. The Impact of Prehabilitation on Patient Outcomes in Hepatobiliary, Colorectal, and Upper Gastrointestinal Cancer Surgery: A PRISMA-Accordant Meta-analysis. Ann Surg. 2021 Jul 1;274(1):70-77. doi: 10.1097/SLA.0000000000004527. PMID 33201129
- See also: study website — http://www.surgicalbridges.co.uk